CLINICAL TRIAL: NCT06880003
Title: Comparison of Cord Blood Preptin Levels in Infants With Low and High Birth Weight for Gestational Age and Infants of Diabetic Mothers With Those of Normal Birth Weight Infants
Brief Title: Cord Blood Preptin Levels in Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Melek Buyukeren, Associate Professor, Konya City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KSH_MB_2025_1
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Newborn Morbidity; Newborn Complication
Keywords: NEWBORN; preptin; UMBİLİCAL CORD BLOOD

STUDY DESIGN:
Intervention Model Description: Between March 2025 and November 2025, mothers of infants born at Konya City Hospital who have either high or low birth weight for their gestational age or are infants of diabetic mothers (study group) will be informed about the study. If they agree to participate, written informed consent will be obtained. Similarly, during the same period, mothers of infants estimated to have normal birth weight for their gestational age (control group) will be informed about the study, and written informed consent will be obtained if they agree to participate.
  Blood samples collected from the umbilical cord at birth will be processed in the biochemistry laboratory, and the serum will be separated and stored at -80°C. After reaching the target sample size, preptin levels will be analyzed. The cost of the kits used for the preptin test will be covered by the researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Appropriate for gestational age (Experimental): During delivery, blood samples will be collected from the umbilical cord of pregnant women who agree to participate in the study.
  Interventions: Other: During delivery, blood samples will be collected from the umbilical cord
- small for gestational age (Experimental): During delivery, blood samples will be collected from the umbilical cord of pregnant women who agree to participate in the study.
  Interventions: Other: During delivery, blood samples will be collected from the umbilical cord
- large for gestational age (Experimental): During delivery, blood samples will be collected from the umbilical cord of pregnant women who agree to participate in the study.
  Interventions: Other: During delivery, blood samples will be collected from the umbilical cord
- Baby of mother diagnosed with GDM (Experimental): During delivery, blood samples will be collected from the umbilical cord of pregnant women who agree to participate in the study.
  Interventions: Other: During delivery, blood samples will be collected from the umbilical cord

INTERVENTIONS:
Other: During delivery, blood samples will be collected from the umbilical cord — During delivery, blood samples will be collected from the umbilical cord of pregnant women who agree to participate in the study.

SUMMARY:
In this study, cord blood preptin levels in infants with high or low birth weight will be compared to those in infants with normal birth weight. Our aim is to determine whether there is a relationship between birth weight and preptin levels. Additionally, we plan to compare the cord blood preptin levels of infants of diabetic mothers with those of normal birth weight infants.

DETAILED DESCRIPTION:
Preptin is the youngest identified member of the insulin family. It is a 34-amino acid protein derived from the E-peptide of pro-insulin-like growth factor 2. Preptin was first isolated in 2001 from the β-cell islet granules of the rat pancreas. It is co-secreted with insulin. In vitro studies have shown that preptin enhances insulin secretion in a dose-dependent manner under high glucose conditions; however, this effect is not observed under normal conditions. Nevertheless, the systemic effects of preptin on glucose metabolism are still not fully understood.

Initial clinical studies have found higher plasma preptin concentrations in patients with type 2 diabetes mellitus compared to individuals with impaired glucose tolerance and healthy controls. Moreover, preptin is linked to insulin resistance by enhancing glucose-mediated insulin secretion. Consequently, elevated preptin levels have been observed in insulin resistance-related conditions such as polycystic ovary syndrome, gestational diabetes, and type 2 diabetes mellitus. In a study serum preptin levels in pregnant women with gestational diabetes were found to be significantly higher than in the control group.

Existing studies on preptin in the literature primarily focus on adults, and there is no comprehensive research on preptin levels in newborns. Based on the available literature, the investigator study aims to compare cord blood preptin levels in infants with high or low birth weight for gestational age and infants of diabetic mothers with those of normal birth weight infants. Through this comparison, The investigators seek to determine whether there is a relationship between preptin levels and an infant's birth weight or the presence of gestational diabetes in the mother.

Between March 2025 and November 2025, mothers of infants born at Konya City Hospital who have either high or low birth weight for their gestational age or are infants of diabetic mothers (study group) will be informed about the study. If they agree to participate, written informed consent will be obtained. Similarly, during the same period, mothers of infants estimated to have normal birth weight for their gestational age (control group) will be informed about the study, and written informed consent will be obtained if they agree to participate.

Blood samples collected from the umbilical cord at birth will be processed in the biochemistry laboratory, and the serum will be separated and stored at -80°C. After reaching the target sample size, preptin levels will be analyzed. The cost of the kits used for the preptin test will be covered by the researchers.

The demographic and clinical characteristics of the patients, as well as prenatal and postnatal risk factors, will be recorded in a patient data collection form. In the investigator's study, preptin levels will be examined in infants of diabetic mothers, infants with high birth weight from healthy mothers, normal birth weight infants, and infants with low birth weight for their gestational age.

No invasive procedures or additional blood sampling will be performed on the patients for the study. The blood samples used will be obtained from residual umbilical cord blood collected for routine tests such as blood gas analysis and blood typing.

ELIGIBILITY:
Inclusion Criteria:

* Large-for-Gestational-Age (LGA) Infants
* Appropriate-for-Gestational-Age (AGA) Infants
* Small-for-Gestational-Age (SGA) Infants
* Infants of Diabetic Mothers (IDM)

Exclusion Criteria:

* Infants with a syndromic appearance or any accompanying disease
* Infants whose families did not provide consent

Ages: 1 Minute to 5 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
serum preptin level | postnatal 5 minutes
  The primary outcome variable is the comparison of serum preptin levels between large-for-gestational-age infants and infants of diabetic mothers with those of normal birth weight infants.The other variable is the comparison of serum preptin levels in small-for-gestational-age infants based on gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: MELEK BUYUKEREN, Principal Investigator — Konya City Hospital
Locations (1):
- Melek Buyukeren, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Once the study is published as a scientific article, it can be shared.

REFERENCES:
- [Background] Ungureanu MC, Bilha SC, Hogas M, Velicescu C, Leustean L, Teodoriu LC, Preda C. Preptin: A New Bone Metabolic Parameter? Metabolites. 2023 Sep 4;13(9):991. doi: 10.3390/metabo13090991. PMID 37755271
- [Background] Aydin S. Three new players in energy regulation: preptin, adropin and irisin. Peptides. 2014 Jun;56:94-110. doi: 10.1016/j.peptides.2014.03.021. Epub 2014 Apr 8. PMID 24721335
- [Background] Buchanan CM, Phillips AR, Cooper GJ. Preptin derived from proinsulin-like growth factor II (proIGF-II) is secreted from pancreatic islet beta-cells and enhances insulin secretion. Biochem J. 2001 Dec 1;360(Pt 2):431-9. doi: 10.1042/0264-6021:3600431. PMID 11716772
- [Background] Cheng KC, Li YX, Asakawa A, Ushikai M, Kato I, Sato Y, Cheng JT, Inui A. Characterization of preptin-induced insulin secretion in pancreatic beta-cells. J Endocrinol. 2012 Oct;215(1):43-9. doi: 10.1530/JOE-12-0176. Epub 2012 Jul 11. PMID 22787110
- [Background] Yang G, Li L, Chen W, Liu H, Boden G, Li K. Circulating preptin levels in normal, impaired glucose tolerance, and type 2 diabetic subjects. Ann Med. 2009;41(1):52-6. doi: 10.1080/07853890802244142. PMID 18618352
- [Background] Celik O, Celik N, Hascalik S, Sahin I, Aydin S, Ozerol E. An appraisal of serum preptin levels in PCOS. Fertil Steril. 2011 Jan;95(1):314-6. doi: 10.1016/j.fertnstert.2010.08.058. PMID 20883990
- [Background] Aslan M, Celik O, Karsavuran N, Celik N, Dogan DG, Botan E, Kafkasli A. Maternal serum and cord blood preptin levels in gestational diabetes mellitus. J Perinatol. 2011 May;31(5):350-5. doi: 10.1038/jp.2010.125. Epub 2010 Dec 16. PMID 21164426
- [Background] Kirac UI, Demir E, Ozkan H, Sahtiyanci B, Uzun H, Ekinci I, Buyukkaba M, Durmus S, Akarsu M, Gelisgen R, Tabak O. Maternal serum preptin levels in the pathogenesis and diagnosis of Gestational diabetes mellitus. J Med Biochem. 2023 Mar 15;42(2):311-317. doi: 10.5937/jomb0-36287. PMID 36987416